CLINICAL TRIAL: NCT06150378
Title: Comparison Between Platelet Rich Plasma and Corticosteroids for the Treatment of Rotator Cuff Tendinopathy Randomized Controlled Double Blind Clinical Trial
Brief Title: Comparison Between Platelet Rich Plasma and Corticosteroids for the Treatment of Rotator Cuff Tendinopathy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital Italiano de Buenos Aires (Other)
Responsible Party: Principal Investigator, LUCIANO ANDRES ROSSI, Shoulder surgeon attending, Clinical professor, Principal investigator, Hospital Italiano de Buenos Aires
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 00005269
Record Dates: First submitted 2023-09-01; First posted 2023-11-29 (Actual); Last update posted 2023-11-29 (Actual); Status verified 2023-11

CONDITIONS: Shoulder Tendinopaty
MeSH Terms: interventions — Adrenal Cortex Hormones

STUDY DESIGN:
Intervention Model Description: Randomized Controlled Double Blind Clinical Trial
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: At the time of blood collection, patients will be placed in a hemotherapy extraction chair with a screen that will prevent the patient from seeing their arm at the time of blood collection.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Corticoid (Active Comparator): Patients that recieve corticosterone injection instead of plathet rich plasma.
  Interventions: Drug: Corticosteroid
- Plathet rich plasma (Experimental): Patients that recieve plathet rich plasma instead of corticoesterone
  Interventions: Biological: Plathet rich plasma

INTERVENTIONS:
Drug: Corticosteroid — Patients that receive an injection with corticosteroid
  Arms: Corticoid
Biological: Plathet rich plasma — Patients that receive an injection with Plathet-rich plasma
  Arms: Plathet rich plasma

SUMMARY:
The goal of this clinical trial is to test if Plateth-rich plasma would provide improved pain relief and function in patients with rotator cuff tendinopathy compared to standard treatment of corticosterone injections.

Researchers will compare a control group of patients treated with a corticosterone injection with a case group of patients treated with Plateth-rich plasma injection.

The purpose of this study is to perform a double-blind randomized controlled trial, comparing PRP with corticosteroids to provide pain relief and improve function in patients with rotator cuff tendinopathy. The hypothesis of this study is that PRP would provide improved pain relief and function in patients with rotator cuff tendinopathy compared to standard treatment of CS injections.

DETAILED DESCRIPTION:
Rotator cuff tendinopathy represents the most common pathology of the shoulder and is the main reason for outpatient consultation for pathologies related to the shoulder girdle. First-line treatment for rotator cuff tendinopathy usually consists of activity modification, stretching and strengthening exercises, oral anti-inflammatory medications. When these initial measures are not effective, a second line of treatment consists of local infiltrations with corticosteroids. However, most of the studies evaluating the effectiveness of corticosteroids in patients with rotator cuff tendinopathy show that the clinical results are usually short-lived.

In this sense, platelet-rich plasma (PRP) emerges as a promising alternative due to its ability to release pro-regenerative growth factors (FsC) and cytokines at the lesion site. Platelet Rich Plasma is considered a minimal handling product. Specifically, at the Hospital Italiano de Buenos Aires (HIBA), platelet-rich plasma has been used for more than 10 years for different musculoskeletal conditions, both on an outpatient basis or as an adjuvant to different surgical procedures.

Several small cohort studies and randomized controlled trials have examined the clinical benefit of PRP for treating patients with rotator cuff tendinopathy, however their results have been confounded by small patient samples, lack of a control group, variable or insufficient data from the PRP preparations and short-term follow-up.

The purpose of this study is to perform a double-blind randomized controlled trial, comparing PRP with corticosteroids to provide pain relief and improve function in patients with rotator cuff tendinopathy. The hypothesis of this study is that PRP would provide improved pain relief and function in patients with rotator cuff tendinopathy compared to standard treatment of CS injections.

Hypothesis

In patients with rotator cuff tendinopathy, PRP subacromial injections produce significantly greater improvement in shoulder pain and function than standard treatment with corticosteroid subacromial injection.

Primary objective To evaluate in patients with rotator cuff tendinopathy whether a subacromial infiltration with PRP produces a significant improvement in pain (measured through the visual analogue scale (VAS) for pain) compared to a control group treated with standard corticosteroid therapy.

Secondary objective To assess whether the use of PRP applied as a subacromial infiltration in patients with rotator cuff tendinopathy improves the functional results (measured using the American Shoulder and Elbow Surgeons (ASES) score) and Constant's score, compared to a control group that underwent subacromial infiltration with corticosteroids.

To assess whether the use of PRP applied as a subacromial infiltration in patients with rotator cuff tendinopathy improves sleep disorders (measured using the Pittsburgh score) compared to a control group that underwent subacromial infiltration with corticosteroids.

Confirm that platelet-rich plasma is a procedure safe by systematically recording adverse effects and complications associated with its use.

To accomplish the objectives, a randomized controlled clinical trial will be conducted, with an intervention group (patients that will receive PRP) and control group (patients that will receive corticosterone), usual treatment, blind for the treatment received by the patient and for clinical and radiological evaluation. The entire study will be carried out at the Hospital Italiano de Buenos Aires headquarters.

Eligible patients will be enrolled in the study by giving their informed consent.

Preparation of platelet-rich plasma

For the PRP group, a leukocyte-poor preparation from a prepackaged kit (RegenLab, Lausanne, Switzerland) will be used. According to the manufacturer's manual, 10 ml of venous blood will be drawn into a blood collection tube containing a sodium citrate anticoagulant and a proprietary separating gel (thixotropic gel) to isolate the red and white blood cells from the PRP. Samples will be centrifuged at 1500g for 5 minutes to produce approximately 7 mL of 80% platelets at 1.6x concentration. The manufacturer reports a filtration of 99.7%, 87 to 89%, 70 to 75%, and 96.5% of red blood cells, white blood cells, mononuclear cells, and granulocytes, respectively. The supernatant is then resuspended by inverting the tube several times and withdrawn into a separate 5 mL syringe for subacromial injection.

This procedure will be performed 2 times in each patient. The product from the first kit will be injected into the patient. Instead, the product from the second kit will be used to evaluate the final composition of the PRP. These specific measurements will include the final average of platelets, leukocytes and erythrocytes, and the specific formula of leukocytes and growth factors.

Statistical analysis raised Quantitative variables will be presented as mean and standard deviation or median and interquartile interval according to the observed distribution. Categorical variables will be presented as proportions. The 95% confidence intervals will be calculated for each of the estimators.

The comparison of continuous data between two groups will be analyzed with the t test if the distribution of the variables is normal or with the Mann-Withney-Wilcoxon test if it is not. The analysis of categorical data will be carried out with the chi-square test. Statistical analysis will be performed with STATA MP version 16 (Stata Corporation, College Station, TX). A p value less than 0.05 will be considered statistically significant.

Sample size To calculate the sample size, the expected values of the variable "pain" represented by the VAS, which is the main outcome variable, are used. The minimal clinically relevant difference (MCID) was previously described in the setting of rotator cuff disease as 1.5 points with a standard deviation of 2.41 points on a 10-point scale for shoulder pain. A type I error probability of 5% and a power of 90% will be used. Using these parameters in a superiority formula, a sample size of 45 patients per group was calculated. Considering the possibility of a loss to follow-up of 10% of the patients per group, 50 patients per group will be included, with a total final sample of 100 patients.

Randomization

All included patients will be randomized after obtaining informed consent. Each patient will be randomly assigned a treatment arm using the online randomizer (http://protocolos.hospitalitaliano.org.ar) to treatment arms 1 (control) or 2 (intervention)

Ethical considerations

Participation in the study will be in all cases voluntary and certified by the informed consent process. The study will be carried out in full accordance with current national and international regulations: Declaration of Helsinki of the World Medical Association, Provision 6677/10 of ANMAT, and the Standards of Good Clinical Practices ICH E6.

The proposed intervention does not frequently present adverse events and there are known contraindications for its application. The procedure will be paid for by the financing of the study, it will not imply any cost to the patient or their health coverage. The costs of monitoring and periodic evaluations will be borne by the study investigators.

All study data will be treated with the utmost confidentiality, with restricted access only to authorized personnel for the purposes of the study in accordance with current legal regulations National Law on Protection of Personal Data 25,326 (Habeas Data Law.

Damage or complications

The coverage for the risk of Institutional Malpractice is attached, of the Clinical Trial that will be contracted to carry out the following study once approved by the Ethics Committee. In the same Coverage is granted to the claim or claims that occur due to any injury, illness or death of Patients, caused or alleged to have been caused by the administration of medicinal products indicated in the Investigation Protocol, by acts of Medical Praxis committed during the execution of the Clinical Trial (negligence, incompetence, imprudence and non-observance of duties). In this multidisciplinary work, 2 Orthopedics and Hemotherapy services will be included. Each service will be responsible for the costs of interventions free of charge and with overtime.

In the case of the preparation of the PRP, will be carried out free of charge and the person in charge will be Dr. Pablo Camino Hemotherapy service plant doctor.

Luciano Rossi doctor of the Shoulder Pathology team of the Orthopedics and Traumatology Service of the Italian Hospital of Buenos Aires will carry out the infiltrations The rehabilitation will be carried out with the standard HIBA kinesiology protocol for patients with chronic rotator cuff tendinopathy and will be carried out by the rehabilitation team of the HIBA Kinesiology service.

ELIGIBILITY:
Inclusion Criteria:

* symptomatic rotator cuff tendinopathy (confirmed by ultrasound).
* At least 3 months of failed conservative treatment (decreased activity, anti-inflammatories, kinesiology for at least 3 months before diagnosis).

Exclusion Criteria:

* Refusal to participate or informed consent
* Previous shoulder surgery,
* Partial or total tears of the rotator cuff,
* Patients with shoulder osteoarthritis
* Advanced fatty infiltration of the rotator cuff muscles
* Systemic or rheumatoid arthritis,
* Uncontrolled diabetes,
* Acute or chronic infections of the shoulder to be operated on
* Ongoing cancer chemotherapy therapies
* Sepsis, septic arthritis, osteomyelitis or other ongoing infectious processes;
* Patients with autoimmune diseases;
* Pregnants

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 100 (Actual)
Dates: Start 2022-09-30 (Actual); Primary Completion 2023-08-01 (Actual); Study Completion 2023-08-31 (Actual)

PRIMARY OUTCOMES:
Visual Analogue Scale (VAS) | 1 year
  From 1 (no pain at all) to 10 (worst pain in patient's life)

SECONDARY OUTCOMES:
ASES (American Shoulder and Elbow Surgeons) | 1 year
  from 0 (worst outcome) to 100 (best outcome)
Constant's score | 1 year
  from 0 (worst outcome) to 100 (best outcome)
Pittsburgh Score | 1 year
  from 0 (worst outcome) to 20 (best outcome)

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Italiano de Buenos Aires, Ciudad de Buenos Aires, Buenos Aires, Argentina

IPD SHARING:
Plan to Share IPD: Undecided
I have not considered that yet

REFERENCES:
- [Background] Garving C, Jakob S, Bauer I, Nadjar R, Brunner UH. Impingement Syndrome of the Shoulder. Dtsch Arztebl Int. 2017 Nov 10;114(45):765-776. doi: 10.3238/arztebl.2017.0765. PMID 29202926
- [Background] Rossi LA, Ranalletta M. Subacromial Decompression Is Not Beneficial for the Management of Rotator Cuff Disease. JBJS Rev. 2020 Jan;8(1):e0045. doi: 10.2106/JBJS.RVW.19.00045. PMID 32105242
- [Background] Diercks R, Bron C, Dorrestijn O, Meskers C, Naber R, de Ruiter T, Willems J, Winters J, van der Woude HJ; Dutch Orthopaedic Association. Guideline for diagnosis and treatment of subacromial pain syndrome: a multidisciplinary review by the Dutch Orthopaedic Association. Acta Orthop. 2014 Jun;85(3):314-22. doi: 10.3109/17453674.2014.920991. Epub 2014 May 21. PMID 24847788
- [Background] Gutierrez-Espinoza H, Araya-Quintanilla F, Cereceda-Muriel C, Alvarez-Bueno C, Martinez-Vizcaino V, Cavero-Redondo I. Effect of supervised physiotherapy versus home exercise program in patients with subacromial impingement syndrome: A systematic review and meta-analysis. Phys Ther Sport. 2020 Jan;41:34-42. doi: 10.1016/j.ptsp.2019.11.003. Epub 2019 Nov 6. PMID 31726386
- [Background] Larsson R, Bernhardsson S, Nordeman L. Effects of eccentric exercise in patients with subacromial impingement syndrome: a systematic review and meta-analysis. BMC Musculoskelet Disord. 2019 Oct 14;20(1):446. doi: 10.1186/s12891-019-2796-5. PMID 31610787
- [Background] Takeno K, Glaviano NR, Norte GE, Ingersoll CD. Therapeutic Interventions for Scapular Kinematics and Disability in Patients With Subacromial Impingement: A Systematic Review. J Athl Train. 2019 Mar;54(3):283-295. doi: 10.4085/1062-6050-309-17. Epub 2019 Mar 4. PMID 30829536
- [Background] Lin MT, Chiang CF, Wu CH, Huang YT, Tu YK, Wang TG. Comparative Effectiveness of Injection Therapies in Rotator Cuff Tendinopathy: A Systematic Review, Pairwise and Network Meta-analysis of Randomized Controlled Trials. Arch Phys Med Rehabil. 2019 Feb;100(2):336-349.e15. doi: 10.1016/j.apmr.2018.06.028. Epub 2018 Aug 2. PMID 30076801
- [Background] Rossi LA, Molina Romoli AR, Bertona Altieri BA, Burgos Flor JA, Scordo WE, Elizondo CM. Does platelet-rich plasma decrease time to return to sports in acute muscle tear? A randomized controlled trial. Knee Surg Sports Traumatol Arthrosc. 2017 Oct;25(10):3319-3325. doi: 10.1007/s00167-016-4129-7. Epub 2016 Apr 16. PMID 27085364
- [Background] Rossi LA, Piuzzi NS, Shapiro SA. Glenohumeral Osteoarthritis: The Role for Orthobiologic Therapies: Platelet-Rich Plasma and Cell Therapies. JBJS Rev. 2020 Feb;8(2):e0075. doi: 10.2106/JBJS.RVW.19.00075. PMID 32015271
- [Background] Rossi LA, Murray IR, Chu CR, Muschler GF, Rodeo SA, Piuzzi NS. Classification systems for platelet-rich plasma. Bone Joint J. 2019 Aug;101-B(8):891-896. doi: 10.1302/0301-620X.101B8.BJJ-2019-0037.R1. PMID 31362555
- [Background] Zicaro JP, Yacuzzi C, Losino A, Costa Paz M. Use of Platelet Rich Plasma for the treatment of patellar tendinopathy. AATD Magazine Volume 25 - N°1 - 2018:30-34
- [Background] Nally FJ, Zanotti G, Buttaro MA, Diaz Dilernia F, Mansilla IG, Comba FM, Piccaluga F. THA conversion rate comparing decompression alone, with autologous bone graft or stem cells in osteonecrosis. Hip Int. 2018 Mar;28(2):189-193. doi: 10.5301/hipint.5000552. Epub 2017 Sep 10. PMID 29027191
- [Background] Murray IR, LaPrade RF, Musahl V, Geeslin AG, Zlotnicki JP, Mann BJ, Petrigliano FA. Biologic Treatments for Sports Injuries II Think Tank-Current Concepts, Future Research, and Barriers to Advancement, Part 2: Rotator Cuff. Orthop J Sports Med. 2016 Mar 31;4(3):2325967116636586. doi: 10.1177/2325967116636586. eCollection 2016 Mar. PMID 27099865
- [Background] Wang D, Rodeo SA. Platelet-Rich Plasma in Orthopaedic Surgery: A Critical Analysis Review. JBJS Rev. 2017 Sep;5(9):e7. doi: 10.2106/JBJS.RVW.17.00024. No abstract available. PMID 28953136
- [Background] Sadoghi P, Lohberger B, Aigner B, Kaltenegger H, Friesenbichler J, Wolf M, Sununu T, Leithner A, Vavken P. Effect of platelet-rich plasma on the biologic activity of the human rotator-cuff fibroblasts: A controlled in vitro study. J Orthop Res. 2013 Aug;31(8):1249-53. doi: 10.1002/jor.22360. Epub 2013 Apr 8. PMID 23568511
- [Background] Hurley ET, Hannon CP, Pauzenberger L, Fat DL, Moran CJ, Mullett H. Nonoperative Treatment of Rotator Cuff Disease With Platelet-Rich Plasma: A Systematic Review of Randomized Controlled Trials. Arthroscopy. 2019 May;35(5):1584-1591. doi: 10.1016/j.arthro.2018.10.115. Epub 2019 Apr 15. PMID 31000394
- [Background] Moraes VY, Lenza M, Tamaoki MJ, Faloppa F, Belloti JC. Platelet-rich therapies for musculoskeletal soft tissue injuries. Cochrane Database Syst Rev. 2014 Apr 29;2014(4):CD010071. doi: 10.1002/14651858.CD010071.pub3. PMID 24782334
- [Background] Michener LA, McClure PW, Sennett BJ. American Shoulder and Elbow Surgeons Standardized Shoulder Assessment Form, patient self-report section: reliability, validity, and responsiveness. J Shoulder Elbow Surg. 2002 Nov-Dec;11(6):587-94. doi: 10.1067/mse.2002.127096. PMID 12469084
- [Background] Constant CR, Gerber C, Emery RJ, Sojbjerg JO, Gohlke F, Boileau P. A review of the Constant score: modifications and guidelines for its use. J Shoulder Elbow Surg. 2008 Mar-Apr;17(2):355-61. doi: 10.1016/j.jse.2007.06.022. Epub 2008 Jan 22. No abstract available. PMID 18218327
- [Background] Backhaus J, Junghanns K, Broocks A, Riemann D, Hohagen F. Test-retest reliability and validity of the Pittsburgh Sleep Quality Index in primary insomnia. J Psychosom Res. 2002 Sep;53(3):737-40. doi: 10.1016/s0022-3999(02)00330-6. PMID 12217446
- [Background] Thigpen CA, Shaffer MA, Gaunt BW, Leggin BG, Williams GR, Wilcox RB 3rd. The American Society of Shoulder and Elbow Therapists' consensus statement on rehabilitation following arthroscopic rotator cuff repair. J Shoulder Elbow Surg. 2016 Apr;25(4):521-35. doi: 10.1016/j.jse.2015.12.018. PMID 26995456
- [Background] Tashjian RZ, Deloach J, Porucznik CA, Powell AP. Minimal clinically important differences (MCID) and patient acceptable symptomatic state (PASS) for visual analog scales (VAS) measuring pain in patients treated for rotator cuff disease. J Shoulder Elbow Surg. 2009 Nov-Dec;18(6):927-32. doi: 10.1016/j.jse.2009.03.021. Epub 2009 Jun 16. PMID 19535272
- [Background] Senn S. Review of Fleiss, statistical methods for rates and proportions. Res Synth Methods. 2011 Sep;2(3):221-2. doi: 10.1002/jrsm.50. Epub 2011 Dec 14. No abstract available. PMID 26061787

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2023-10-10): https://cdn.clinicaltrials.gov/large-docs/78/NCT06150378/Prot_SAP_000.pdf
  • Informed Consent Form (2023-10-10): https://cdn.clinicaltrials.gov/large-docs/78/NCT06150378/ICF_001.pdf